CLINICAL TRIAL: NCT00560794
Title: Open-label, Multicenter Phase II Study to Investigate the Efficacy, Safety, and Tolerability of the Bispecific T-cell Engager (BiTE®) MT103 in Patients With Minimal Residual Disease of B-precursor Acute Lymphoblastic Leukemia
Brief Title: Phase II Study of the BiTE® Blinatumomab (MT103) in Patients With Minimal Residual Disease of B-precursor Acute Lymphoblastic Leukemia (ALL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen Research (Munich) GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT103-202; 2006-006520-19 (EudraCT Number)
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2015-01-07 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2014-12

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Minimal Residual Disease; adult ALL; immunotherapeutic treatment; anti-CD19 bispecific antibody derivative; Blinatumomab; MT103
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Neoplasm, Residual | interventions — blinatumomab; N,N-dicyclohexyl-isoborneol-10-sulfonamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blinatumomab (Experimental): Participants received blinatumomab as continuous intravenous infusion at constant flow rate over 4 weeks followed by a 2 week treatment-free period (defined as one treatment cycle), for up to a maximum of 10 cycles. The initial dose was 15 μg/m^2/day. A dose increase to 30 μg/m^2/day was permitted with evidence for insufficient response to blinatumomab treatment.
  Interventions: Biological: Blinatumomab (MT103)

INTERVENTIONS:
Biological: Blinatumomab (MT103) — Administered by continuous intravenous (CIV) over 4 weeks per cycle
  Other Names: Blinatumomab; AMG103; MT103; BLINCYTO™

SUMMARY:
The purpose of this study is to determine whether the bispecific T-cell engager (BiTE®) Blinatumomab (MT103) is effective in the treatment of ALL patients with minimal residual disease.

DETAILED DESCRIPTION:
The presence of leukemia cells below the cytological detection limit (5% leukemic cells) is defined as minimal residual disease (MRD). If no MRD is detectable (< 10^-4 = less than 1 leukemia cell per 10^4 bone marrow cells) a complete molecular remission is reached. In the last years a series of retrospective studies has shown that MRD in adult ALL is an independent prognostic factor as already demonstrated for childhood leukemia. Diagnostic tools for MRD are polymerase chain reaction (PCR) and/or flow cytometry. PCR analysis can detect fusion transcripts such as bcr/abl and individual clonal rearrangements of immunoglobulins (IgH) and/or T-cell receptor genes (TCR). About 25% of patients with MRD defined by rearrangement comprise a high-risk group with a 94% relapse rate within 3 years. In general for patients with MRD, who are not eligible for allogenic stem cell transplantation, curative treatment is not available. This accounts for MRD defined by the Philadelphia chromosome translocation as well as for MRD defined by rearrangement. The current study is set up to address the question of treating MRD positive ALL with the bispecific anti-cluster of differentiation (CD)19 x anti-CD3 antibody derivative blinatumomab (MT103).

ELIGIBILITY:
Inclusion Criteria:

* B-precursor ALL patients in complete hematological remission with molecular failure or molecular relapse starting at any time after consolidation I of front-line therapy within German Multicenter Study Group on Adult Acute Lymphoblastic Leukemia (GMALL) standards or at any time outside GMALL standards.
* Patients must have a molecular marker for evaluation of minimal residual disease which is either Breakpoint cluster region/gene on human chromosome #9 (Bcr/abl) at any detection level or individual rearrangements of immunoglobulin or T-cell receptor (TCR)-genes measured by an assay with a sensitivity of minimum 10^-4: At least one individual marker at a quantitative level ≥ 10^-4.
* Eastern Cooperative Oncology Group (ECOG) Performance Status < 2
* Ability to understand and willingness to sign a written informed consent
* Signed and dated written informed consent is available

Exclusion Criteria:

* Current extra medullar involvement
* History of or current relevant central nervous system (CNS) pathology (except migraine/headache and/or previous infiltration of cerebrospinal fluid (CSF) by ALL)
* Current infiltration of cerebrospinal fluid by ALL
* History of or current autoimmune disease
* Autologous stem cell transplantation within 6 weeks prior to study entry
* Any prior allogeneic stem cell transplantation
* Cancer chemotherapy within 4 weeks prior to study treatment (except for intrathecal prophylaxis and/or low dose maintenance therapy such as vinca alkaloids, mercaptopurine, methotrexate, steroids)
* Radiotherapy within 4 weeks prior to study treatment
* Therapy with monoclonal antibodies (Rituximab, MabCampath) within 6 weeks prior to study treatment
* Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation
* Presence of human anti-murine antibodies (HAMA)
* Abnormal bone marrow, renal or hepatic function
* Indication for a hypercoagulative state
* History of malignancy other than ALL within 5 years prior to study entry, with the exception of basal cell carcinoma of the skin or cervix carcinoma in situ
* Active severe infection, any other concurrent disease or medical condition that are deemed to interfere with the conduct of the study as judged by the investigator
* Known infection with human immunodeficiency virus (HIV) or chronic infection with hepatitis B virus (HbsAg positive) or hepatitis C virus (anti-HCV positive)
* Pregnant or nursing women
* Women of childbearing potential not willing to use an effective form of contraception during participation in the study and at least 3 months thereafter or male patients not willing to ensure effective contraception during participation in the study and at least three months thereafter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Bargou, Professor, Principal Investigator — Julius-Maximilians-Universität Würzburg
Locations (6):
- Germany (6):
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Julius-Maximilians-Universität Würzburg, Würzburg, Bavaria
  - Klinikum der J.W. Goethe Universität, Frankfurt am Main, Hesse
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitätsklinikum Schleswig-Holstein im Städtischen Krankenhaus Kiel, Kiel, Schleswig-Holstein

REFERENCES:
- [Derived] Zhu M, Wu B, Brandl C, Johnson J, Wolf A, Chow A, Doshi S. Blinatumomab, a Bispecific T-cell Engager (BiTE((R))) for CD-19 Targeted Cancer Immunotherapy: Clinical Pharmacology and Its Implications. Clin Pharmacokinet. 2016 Oct;55(10):1271-1288. doi: 10.1007/s40262-016-0405-4. PMID 27209293
- [Derived] Zugmaier G, Topp MS, Alekar S, Viardot A, Horst HA, Neumann S, Stelljes M, Bargou RC, Goebeler M, Wessiepe D, Degenhard E, Gokbuget N, Klinger M. Long-term follow-up of serum immunoglobulin levels in blinatumomab-treated patients with minimal residual disease-positive B-precursor acute lymphoblastic leukemia. Blood Cancer J. 2014 Sep 5;4(9):244. doi: 10.1038/bcj.2014.64. No abstract available. PMID 25192414
- [Derived] Klinger M, Brandl C, Zugmaier G, Hijazi Y, Bargou RC, Topp MS, Gokbuget N, Neumann S, Goebeler M, Viardot A, Stelljes M, Bruggemann M, Hoelzer D, Degenhard E, Nagorsen D, Baeuerle PA, Wolf A, Kufer P. Immunopharmacologic response of patients with B-lineage acute lymphoblastic leukemia to continuous infusion of T cell-engaging CD19/CD3-bispecific BiTE antibody blinatumomab. Blood. 2012 Jun 28;119(26):6226-33. doi: 10.1182/blood-2012-01-400515. Epub 2012 May 16. PMID 22592608

RESULTS

PARTICIPANT FLOW:
Groups:
- Blinatumomab: Participants received blinatumomab as continuous intravenous infusion at constant flow rate over 4 weeks followed by a 2 week treatment-free period (defined as one treatment cycle), for up to a maximum of 10 cycles. The initial dose was 15 μg/m²/day. A dose increase to 30 μg/m²/day was permitted with evidence for insufficient response to blinatumomab treatment.
Period: Overall Study
Arm/Group | Blinatumomab
Started | 21
Completed 1 Treatment Cycle | 20
Completed | 10
Not Completed | 11
Not completed — Adverse Event | 2
Not completed — Patient was not Compliant | 1
Not completed — Minimal Residual Disease Relapse | 1
Not completed — Hematological Relapse | 1
Not completed — Received Bone Marrow Transplant | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants who received ≥ 1 infusion of blinatumomab who completed at least the first treatment cycle and for whom at least one minimal residual disease (MRD) response assessment was available.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.8 (18.3)
Age, Customized [Number; unit: participants]
  20-30 years | 3
  31-40 years | 5
  41-50 years | 2
  51-60 years | 1
  61-70 years | 7
  > 70 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 20
Genetic Alterations [Number; unit: participants] — bcr/abl: breakpoint cluster region; Ig: immunoglobulin; TCR: T-cell receptor. For bcr/abl above detection limit and t(4;11) translocation above detection limit participants may have rearrangements in addition to translocations.
  For Rearrangements of immunoglobulin / TCR genes participants did not show any translocation.
  participants
    bcr/abl translocation above detection limit | 5
    t(4;11) translocation above detection limit | 2
    Rearrangements of Ig / TCR genes only | 13
    Rearrangements of Ig / TCR genes & translocations | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Minimal Residual Disease (MRD) Response Within 4 Cycles of Treatment
Description: MRD Response is defined as:
  * If Philadelphia Chromosome (Ph) positive (+) or translocation (t) (4;11), response was achieved when Ph or t(4;11) was below detection limit and individual rearrangements of immunoglobulin or T-cell receptor genes are below 10^-4.
  * If Ph and t(4;11) negative, response was achieved when individual rearrangements of immunoglobulin or T-cell receptor genes are below 10^-4.
Time Frame: Within 4 treatment cycles, 24 weeks
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 20
percentage of participants | 80.0 [56.3 to 94.3]
Statistical Analysis 1: Comparison: Blinatumomab; Test type: Superiority or Other; p = 0.0000, 1-sided exact binomial test — The null hypothesis stated that the true MRD response probability (π) ≤ 5%

2. Secondary Outcome: Percentage of Participants With an MRD Response After Each Treatment Cycle
Description: MRD Response is defined as:
  * If Philadelphia Chromosome (Ph)+ or t(4;11), response was achieved when Ph or t(4;11) was below detection limit and individual rearrangements of immunoglobulin or T-cell receptor genes are below 10^-4.
  * If Ph and t(4;11) negative, response was achieved when individual rearrangements of immunoglobulin or T-cell receptor genes are below 10^-4.
Time Frame: At the end of each treatment cycle - Weeks 4, 10, 16, and 22.
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 20
percentage of participants
  MRD negativity achieved after cycle 1 | 80.0 [56.3 to 94.3]
  MRD negativity achieved after cycle 2 | 80.0 [56.3 to 94.3]
  MRD negativity achieved after cycle 3 | 80.0 [56.3 to 94.3]
  MRD negativity achieved after cycle 4 | 80.0 [56.3 to 94.3]

3. Secondary Outcome: Time to Hematological Relapse
Description: The time to hematological relapse is defined as the time between start of first infusion of blinatumomab and the first result of hematological relapse. Participants without an event of hematological relapse were censored on their last available date of bone marrow aspiration/biopsy.
  Hematological relapse is defined as > 5% leukemia cells in bone marrow. Time to hematological relapse was analyzed using Kaplan-Meier methods.
Time Frame: Up to the data cut-off date of 14 January 2010; maximum duration of follow-up was 564 days.
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Blinatumomab
Number analyzed (Participants) | 20
days | NA [NA to NA] — The median time to hematological relapse was not reached due to the low number of events

4. Secondary Outcome: Time to MRD Progression
Description: Time to MRD progression is defined for participants who do not show MRD response at any time during the study as the time from start of first infusion until the first result of MRD progression or hematological relapse, if no MRD progression was diagnosed before hematological relapse. For participants who showed MRD response during the study the time to MRD progression is defined as the time from the date of the first MRD response to the date of MRD relapse. Participants without an event of MRD progression were censored on the day of their last bone marrow aspiration/biopsy. Participants who received a bone marrow transplant were censored on the last day of bone marrow aspiration/biopsy before transplantation.
  MRD progression is defined as the increase in the MRD level by 1 log as compared to the baseline level (equal to a 10-fold increase in the number of MRD cells), and had to be confirmed within 6 weeks.
Time Frame: Up to the data cut-off date of 14 January 2010; Median follow-up time was 155 days
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Blinatumomab
Number analyzed (Participants) | 20
days | 221.0 [170.0 to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Time to MRD Relapse
Description: Time to MRD relapse is defined only for participants with an MRD response during the study, defined as the time between the date of the first MRD response and the date of MRD relapse. If a participant experienced hematological relapse without having shown MRD positivity before then the time point of MRD relapse is defined as the time point of hematological relapse. Participants without an event of MRD relapse or hematological relapse were censored on the day of their last available bone marrow aspiration/biopsy. If a participant received a bone marrow transplant the last day of bone marrow aspiration/biopsy before transplantation was used as time point for censoring.
  MRD relapse is defined as reappearance of bcr/abl, and/or t(4;11) translocation at any detection level, and/or by individual rearrangements of immunoglobulin or T-cell receptor genes ≥10^-4 for at least 1 individual marker measured by an assay with a sensitivity of minimum 10^-4 and should be confirmed within 6 weeks.
Time Frame: Up to the data cut-off date of 14 January 2010; Median follow-up time was 116.5 days
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Blinatumomab
Number analyzed (Participants) | 15
days | NA [NA to NA] — Median was not reached during the study due to the low number of events

6. Secondary Outcome: Number of Participants With Adverse Events
Description: The severity (or intensity) of AEs was evaluated according to the grading scale provided in the Cancer Therapy Evaluation Program, Common Terminology Criteria for Adverse Events (CTCAE), version 3.0, or according to the following: Grade 1 - Mild AE; Grade 2 - Moderate AE; Grade 3 - Severe AE; Grade 4 - Life-threatening or disabling AE; Grade 5 - Death.
  The investigator used medical judgment to determine if there was a causal relationship (ie, related, unrelated) between an adverse event and blinatumomab.
  A serious adverse event (SAE) is any untoward medical occurrence or effect that, at any dose results in death, is life-threatening, requires or prolongs hospitalization, results in persistent or significant disability or incapacity, or is a congenital anomaly or birth defect. In addition, all laboratory abnormalities of grade four severity that occur during or after administration of the investigational drug, any overdose and a pregnancy or fathering were reported as SAEs.
Time Frame: From the start of study treatment until up to 4 weeks after the end of study treatment. The median treatment duration was 87.3 days.
Population: Safety analysis set, including all participants who received ≥ 1 infusion of blinatumomab.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 21
participants
  Any adverse event | 21
  Adverse events of at least CTC grade 3 | 17
  Treatment-related adverse events | 21
  Related adverse events of at least CTC grade 3 | 13
  Serious adverse evets | 10
  Related serious adverse events | 9
  AEs leading to discontinuation of blinatumomab | 1
  AEs leading to death | 0

7. Secondary Outcome: Change From Screening Value in B-cell Count During Cycle 1
Description: B-cells were measured by flow cytometry.
Time Frame: At Screening and in Cycle 1 at the start of infusion, 45 minutes, 2, 6, 12, 24 hours and at Days 2, 7, 14, 21, 28 and 35 after the start of infusion.
Population: Participants who received blinatumomab with available pharmacodynamic data.
Measure: Mean (Standard Deviation); unit: cells/μL
Groups:
- Blinatumomab: Participants received blinatumomab 15 μg/m²/day as continuous intravenous infusion at constant flow rate over 4 weeks followed by a 2 week treatment-free period.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 19
cells/μL
  Start of infusion (N=19) | 0.0181 (0.0803)
  45 minutes (N=19) | -0.0098 (0.0402)
  2 hours (N=18) | -0.0361 (0.0621)
  6 hours (N=19) | -0.0435 (0.0685)
  12 hours (N=16) | -0.0417 (0.0689)
  24 hours (N=18) | -0.0403 (0.0700)
  Day 2 (N=17) | -0.0310 (0.0589)
  Day 7 (N=18) | -0.0462 (0.0717)
  Day 14 (N=18) | -0.0490 (0.0745)
  Day 21 (N=18) | -0.0494 (0.0747)
  Day 28 (N=17) | -0.0392 (0.0634)
  Day 35 (N=18) | -0.0493 (0.0748)

8. Secondary Outcome: Change From Screening Value in T-cell Count During Cycle 1
Description: T-cells were measured by flow cytometry.
Time Frame: as for outcome 7
Population: Participants who received blinatumomab with available pharmacodynamic data.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 19
cells/μL
  Start of infusion (N=19) | -0.0418 (0.2925)
  45 minutes (N=19) | -0.3208 (0.3137)
  2 hours (N=18) | -0.4976 (0.3454)
  6 hours (N=19) | -0.5227 (0.3432)
  12 hours (N=16) | -0.5390 (0.3649)
  24 hours (N=18) | -0.4780 (0.3774)
  Day 2 (N=17) | -0.3328 (0.3704)
  Day 7 (N=18) | 0.1231 (0.3051)
  Day 14 (N=18) | 0.1172 (0.4671)
  Day 21 (N=18) | 0.1975 (0.5596)
  Day 28 (N=17) | 0.1687 (0.3119)
  Day 35 (N=18) | 0.2271 (0.3739)

9. Secondary Outcome: Serum Cytokine Peak Levels in Cycle 1
Description: The activation of immune effector cells was monitored by the measurement of peripheral blood cytokine levels including interleukin (IL)-2, IL-4, IL-6, IL-8, IL-10, tumor necrosis factor (TNF)-α and interferon gamma (IFN)-γ using fluorescence-activated cell sorter (FACS)-based cytometric bead array (CBA) system.The limit of detection (LOD) for the cytokine determination was 20 pg/mL, the limit of quantification (LOQ) was 125 pg/mL.
Time Frame: Cycle 1 at pre-dose and at post infusion start at 45 minutes; 2, 6, 12, 24, and 48 hours; 7, 14, 21, and 28 days.
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Blinatumomab: Participants received blinatumomab 15 μg/m²/day as continuous intravenous infusion at constant flow rate over 4 weeks.
Arm/Group | Blinatumomab
Number analyzed (Participants) | 21
pg/mL
  IL-2 | NA (NA) — Levels less than the limit of quantitation
  IL-4 | NA (NA) — Levels less than the limit of detection
  IL-6 | 693.2 (1122.9)
  IL-8 | NA (NA) — Levels less than the limit of detection
  IL-10 | 1135.3 (1155.6)
  IFN-γ | 408.5 (614.3)
  TNF-α | NA (NA) — Levels less than the limit of quantitation

10. Secondary Outcome: Serum Blinatumomab Concentration at Steady State
Description: The mean serum concentration of blinatumomab during cycle 1. The LOQ of the assay was 100 pg/mL, and the limit of detection (LOD) was 3 pg/mL.
Time Frame: Cycle 1 at predose and at 2, 6, and 12 hours after start of infusion then weekly until end of the cycle, and at 1, 2, 4, 6, 8, and 24 hours after stop of infusion.
Population: Participants who received at least 1 infusion of blinatumomab with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 19
pg/mL | 696 (147)

11. Secondary Outcome: Area Under the Drug Concentration-time Curve From Time Zero to Infinity
Time Frame: as for outcome 10
Population: Participants who received at least 1 infusion of blinatumomab with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Blinatumomab
Number analyzed (Participants) | 18
hr*ng/mL | 481 (106)

12. Secondary Outcome: Apparent Volume of Distribution
Time Frame: as for outcome 10
Population: Participants who received at least 1 infusion of blinatumomab with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: L/m²
Arm/Group | Blinatumomab
Number analyzed (Participants) | 18
L/m² | 2.00 (0.95)

13. Secondary Outcome: Clearance of Blinatumomab
Time Frame: as for outcome 10
Population: Participants who received at least 1 infusion of blinatumomab with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: L/hr/m²
Arm/Group | Blinatumomab
Number analyzed (Participants) | 19
L/hr/m² | 0.939 (0.199)

14. Secondary Outcome: Terminal Half-life of Blinatumomab
Time Frame: as for outcome 10
Population: Participants who received at least 1 infusion of blinatumomab with available pharmacokinetic data.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Blinatumomab
Number analyzed (Participants) | 18
hours | 1.47 (0.53)

ADVERSE EVENTS:
Time Frame: From the start of study treatment until up to 4 weeks after the end of study treatment. The median treatment duration was 87.3 days.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
  Summary of Adverse Events includes only those participants who received at least one dose of investigational product.
Arm/Group | Blinatumomab
Serious Adverse Events (participants affected / at risk) | 10/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=21)
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Bacterial sepsis (Infections and infestations) | 1
Bronchopneumonia (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Escherichia sepsis (Infections and infestations) | 1
Medical device complication (Injury, poisoning and procedural complications) | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 1
Convulsion (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Blinatumomab (N=21)
Leukopenia (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Bradycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 4
Lacrimation increased (Eye disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 3
Catheter site erythema (General disorders) | 2
Catheter site pain (General disorders) | 2
Chills (General disorders) | 9
Fatigue (General disorders) | 8
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 21
Immunodeficiency (Immune system disorders) | 2
Bronchitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Oral herpes (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 4
Blood alkaline phosphatase increased (Investigations) | 2
Blood immunoglobulin A decreased (Investigations) | 14
Blood immunoglobulin G decreased (Investigations) | 13
Blood immunoglobulin M decreased (Investigations) | 10
Blood lactate dehydrogenase increased (Investigations) | 2
Blood potassium decreased (Investigations) | 3
C-reactive protein increased (Investigations) | 6
Coagulation factor XIII level increased (Investigations) | 2
Fibrin D dimer increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 5
Immunoglobulins decreased (Investigations) | 2
Monocyte count increased (Investigations) | 2
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 6
Growing pains (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 10
Tremor (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 5
Haematuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Night sweats (Skin and subcutaneous tissue disorders) | 2
Periorbital oedema (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 2
Hypotension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.